CLINICAL TRIAL: NCT05950022
Title: Study Evaluating the Clinical Improvement Obtained by Endoscopic Tenotomy of the Ilio-Psoas, at the Level of the Lesser Trochanter Versus at the Level of the Acetabular Notch, on Psoas Cup Impingements After Total Hip Prosthesis
Brief Title: Clinical Improvement Obtained by Endoscopic Ilio-Psoas Tenotomy (Lesser Trochanter Versus Acetabular Notch)
Acronym: ETIPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A00802-43
Record Dates: First submitted 2023-07-04; First posted 2023-07-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: Interventional, comparative, randomized study, in 2 parallel groups, single-blind
Who Masked: Participant
Masking Description: The patient does not know which technique he will benefit from, the surgeon will proceed with the surgery and will therefore be informed of the result of the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic tenotomy at the level of the lesser trochanter (Experimental): Patients will benefit from endoscopic tenotomy surgery of the iliopsoas tendon at the level of the lesser trochanter.
  Interventions: Procedure: Endoscopic tenotomy surgery of the iliopsoas tendon
- Endoscopic tenotomy at the level of the acetabular notch (Experimental): Patients will benefit from endoscopic tenotomy surgery of the iliopsoas tendon at the level of the acetabular notch.
  Interventions: Procedure: Endoscopic tenotomy surgery of the iliopsoas tendon

INTERVENTIONS:
Procedure: Endoscopic tenotomy surgery of the iliopsoas tendon — The surgery will be performed under general anesthesia with standardized multimodal analgesia. Whatever the techniques, the approaches, the instruments to perform the procedure and the postoperative course will be identical, as in usual practice.

SUMMARY:
The purpose of the study is to assess Oxford Hip Score at baseline, at 2 months and at over 12 months.

DETAILED DESCRIPTION:
This is an interventional, comparative, randomized study, in 2 parallel groups, single-blind (the patient does not know which technique he will benefit from, the surgeon will carry out the surgery and will therefore be informed of the result of the randomization ) and monocentric.

Comparative prospective cohort study of an endoscopic tenotomy surgery of the iliopsoas tendon at the level of the lesser trochanter versus at the level of the acetabular notch, in the context of anterior pain for impingement between the iliopsoas tendon and the prosthetic cup in patients after Total Hip Prosthesis.

The study will be proposed to the patient during the preoperative consultation. Patients eligible for surgery will be offered the study. After a reflection period of at least 15 days, patients who agree to participate in the study will be included. Randomization will be done by drawing lots to decide whether the endoscopic tenotomy will be performed at the level of the lesser trochanter or at the level of the acetabular notch. The surgery will be performed under general anesthesia with standardized multimodal analgesia. Whatever the techniques, the approaches, the instruments to perform the procedure and the postoperative course will be identical, as in usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Definite diagnosis of iliopsoas tendinopathy due to conflict between the tendon and the prosthetic cup;
* Failure of first-line conservative treatment;
* Planned endoscopic tenotomy;
* Affiliation to the social security scheme;
* Signed informed consent.

Exclusion Criteria:

* Revision total hip prosthesis, multiple operations prior to tenotomy;
* Other surgical or medical interventions planned during the study;
* Participation in another clinical trial, or during a period of exclusion from another clinical trial;
* Pregnant or likely to be pregnant (of childbearing age, without effective contraception) or breastfeeding;
* Patient deprived of liberty or under guardianship or curatorship or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score | 1 year
  Compare the clinical improvement experienced by patients having an endoscopic tenotomy of the iliopsoas tendon at the level of the lesser trochanter versus at the level of the notch at more than 1 year minimum.
  The Oxford Hip Score is a self-administered patient-administered 12-item "Patient Reported Outcome Measures" questionnaire that allows the surgeon to assess clinical outcomes after total hip replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No